CLINICAL TRIAL: NCT07240636
Title: Study of Food Effects of VV119 Capsules in Chinese Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VV119-03
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): Subjects will receive VV119 orally for single dose.
  Interventions: Drug: VV119
- B group (Experimental): Subjects will receive VV119 orally for single dose.
  Interventions: Drug: VV119

INTERVENTIONS:
Drug: VV119 — A：2 mg VV119, following an overnight fast of at least 10 hours for Period 1; 2mg VV119, administered 30 minutes after the start of a Standard meal for Period 2;
  Arms: A group
Drug: VV119 — B: 2mg VV119, administered 30 minutes after the start of a Standard meal for Period 1;2mg VV119, following an overnight fast of at least 10 hours for Period 2；
  Arms: B group

SUMMARY:
This study is a single-center, randomized, open label, 2×2 crossover design to assess the standard meal effects on PK of a single oral dose of VV119 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males:aged 18 to 45 years old, males ,Body weight no less than 50.0 kg ; females :Aged 18 to 60 years old ,Body weight no less than 45.0 kg ,Body Mass Index of 19.0 to 26.0kg/m2,
2. Medically healthy, Physical examination, vital signs examination, laboratory examination, electrocardiogram examination results were normal or abnormal without clinical significance,
3. Males subjects who are willing to take effective contraceptive during the study and within 3 months after the study completed; females not of child-bearing potential,
4. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. With current or past medical history diseases or dysfunction that affect the clinical trial, evaluated by the investigator, including but not limited to central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, blood system, ophthalmology and other diseases, history of malignant tumor or other diseases that are not suitable for participating in the clinical trial;
2. With current or previous mental disorders and brain dysfunction, or suicide risk according to the clinical judgment of the investigator, or a history of self-mutilation;
3. With any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial, such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, history of gastrointestinal bleeding, etc.
4. With a known history of allergy to investigating drug ingredients or similar drugs, a history of allergic diseases or allergic constitution;
5. Positive for hepatitis B virus surface antigen (HBsAg), or syphilis antibody (Anti-TP), or hepatitis C antibody (anti-HCV), or human immunodeficiency virus antigen/antibody combined detection (HIV-Ag/Ab);
6. With a history of surgery within 3 months before screening, or have not recovered from surgery, or have an expected surgical plan during the trial;
7. With a blood donation or blood loss ≥ 400 mL within 3 months before screening, or a blood donation or blood loss ≥ 200 mL within 1 month, or a history of blood product use within 3 months before screening;
8. Taking any prescription drugs, over-the-counter drugs, and any functional vitamins or herbal products within 2 weeks before screening;
9. Using any drugs that inhibit or induce hepatic drug metabolizing enzymes CYP3A4, CYP3A5, CYP2D6 (such as inducers - phenobarbital, rifampicin, carbamazepine, phenytoin sodium, glucocorticoids, etc.; inhibitors - ketoconazole, itraconazole, cimetidine, clarithromycin, verapamil, erythromycin, etc.) within 4 weeks (or 5 half-lives, whichever is longer) before screening;
10. Participating in any clinical trial and taking clinical trial drugs within 3 months before screening, or being participating in other clinical trials;
11. Smoke test positive or smoking more than 5 cigarettes per day or average intake of coffee or tea more than 5 cups per day (200 mL/cup) within 3 months before screening, or unable to stop users during the study;
12. With alcohol abuse within 1 year before screening, average weekly alcohol intake more than 14 standard units [1 unit = 360 mL beer (alcohol content 5%) or 45 mL spirits (alcohol content 40%) or 150 mL wine (alcohol content 12%)] or positive for alcohol breath test;
13. With a history of drug abuse within 1 year before screening, or positive for urine drug screening;
14. With a family history of sudden cardiac death (sudden death age less than 40 years);
15. With a resting pulse < 50 beats/min or ≥ 100 beats/min; resting systolic blood pressure < 85 mmHg or ≥ 140 mmHg; resting diastolic blood pressure < 50 mmHg or ≥ 90 mmHg; systolic blood pressure decreased by ≥ 20 mmHg and/or diastolic blood pressure decreased by ≥ 10 mmHg and/or accompanied by clinical symptoms within 3 minutes of standing;
16. Abnormal in 12-lead electrocardiogram (ECG), clinically significant judged by the investigator (e.g., QTcF> 450 ms in men and > 470 ms in women);
17. With the aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine (Cr), urea (Urea), serum prolactin levels beyond the upper limit of normal (ULN);
18. Having special requirements for food, unable to observe a unified diet or having dysphagia;
19. Rejecting abide by the following conditions during the trial: smoking, alcohol or caffeine-containing beverages are prohibited, and strenuous exercise is avoided;
20. Directly related to this clinical trial;
21. Other subjects that the investigator considers inappropriate for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Dosing through follow-up call (7 days after last dose of investigational product)
  Incidence of Treatment-Emergent Adverse Events
Cmax | 480 hours after dosing
  maximum observed plasma concentration of the main metabolites VV119-M2
AUC0-∞ | 480 hours after dosing
  area under the plasma concentration time curve from time zero to infinity of the main metabolites VV119-M2
AUC0-t | 480 hours after dosing
  area under the plasma concentration time curve from time zero to the last of the main metabolites VV119-M2

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No